CLINICAL TRIAL: NCT03834857
Title: Stentrode With Thought-controlled Digital Switch: An Early Feasibility Study (EFS) of the Safety of the Stentrode Device in Participants With Loss of Motor Function Due to Paralysis
Brief Title: SWITCH: Stentrode First-in-Human Study of Implantable BCI for Control of a Digital Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synchron Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Synchron, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S-01-01
Record Dates: First submitted 2019-02-01; First posted 2019-02-08 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Insertion of Stentrode TM device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single (Other): Implantation of Stentrode device
  Interventions: Device: Stentrode

INTERVENTIONS:
Device: Stentrode — Implantation of Stentrode device

SUMMARY:
SWITCH Study

DETAILED DESCRIPTION:
STENTRODE WITH THOUGHT CONTROLLED DIGITAL SWITCH: An early feasibility study (EFS) of the safety of the StentrodeTM device in participants with loss of motor function due to paralysis from spinal cord injury, motor neuron disease, stroke, muscular dystrophy or loss of limbs.

Research has shown that in individuals with neurological conditions, brain signals can be recorded using electrical sensors implanted on to the brain. These signals could be used by the individuals to control assistive technology (e.g. spelling devices) that help with daily life, just by thinking. However, implanting these electrical sensors often requires open brain surgery.

A new medical device and surgical technique has been developed, which allows implantation of the electrical sensors without open brain surgery. The device, called Stentrode™, is a small metallic mesh tube (stent), with electrode contacts (small metal disks) within the stent structure. It can be placed inside a blood vessel of the brain located in the motor cortex. This does not involve open brain surgery.

The purpose of this research is to evaluate the safety of the Stentrode™ device in humans. This is an experimental device. This research will be the first of its kind to be performed in humans and may help find safer, more effective ways to introduce/implant electrical sensors in patients. This could foster the development of user friendly biotechnology for patients with neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of spinal cord injury (SCI), motor neurone disease (MND) [also known as amyotrophic lateral sclerosis (ALS)], stroke, muscular dystrophy or loss of limbs.
2. Diagnosed for at least six (6) months and if SCI, at least twelve (12) months
3. Aged between 18 and 75 years of age; females must be of non-child bearing potential or with negative pregnancy test and not breast feeding
4. Life expectancy of at least twelve (12) months in the opinion of the treating physician
5. Understands English
6. Is computer literate
7. Is willing and able to access all clinical testing locations and is not impeded by geographical location (ie: ideally lives within 100 kms or Less than 2 hours travel time to study site)
8. No conditions, including an eye movement disorder, that would prevent the use of eye tracking software and has a level of vision that will not impede viewing of screens and visualisations
9. Has normal venous sinus anatomy, with two patent jugular veins (of sufficient size for the device) and bilateral patent transverse sinuses as evidenced by MR venography (MRV) or CT venography (CTV) within the last six (6) months or if vascular anatomy is unknown, is willing to undergo an MRV or CTV assessment to assess vascular suitability for endovascular device placement
10. Evidence of activation, under fMRI testing, of motor cortical areas adjacent to the superior sagittal sinus

Exclusion Criteria:

1. Is unwilling to comply with all procedures relating to study
2. Based on the doctors opinion, has unrealistic expectations regarding the possible benefits, risks and limitations associated with the implantation or surgical procedures
3. Has dementia or cognitive impairment sufficient to impair capacity to provide informed consent or which could impact ability to comply with investigational requirements (eg: MMSE <24, ECAS or other determination made by Investigator)
4. For MND participants, has NOT had a formal capacity assessment by a professional with experience in capacity assessment (psychiatrist, neurologist, psychologist) within 90 days of Screen1 visit, which assesses capacity to consent and excludes Frontotemporal dementia
5. Has a history of substance abuse within the preceding two (2) years
6. Chronic oral or intravenous steroids or immunosuppressive therapy or other therapy/clinical condition that severely reduces immunity Has been hospitalized for a psychiatric condition with the preceding two (2) years or has had a history of psychosis within the preceding two (2) years
7. Has a contraindication to magnetic resonance imaging (MRI)
8. Has an active implanted stimulation device (eg: pacemaker, deep brain stimulator, spinal cord stimulator)
9. Is deemed unsuitable by a specialist anaesthesiologist or respiratory physician to undergo a general anaesthetic
10. Has findings on MRV deemed incompatible, by an experienced neurointerventionalist, with device implantation in the SSS [eg: isolated dominant, superior anastomotic vein (vein of Trolard)]
11. Has a contraindication to angiographic imaging, including chronic kidney injury (CKI -eGFR < 60mls/min)
12. Has known allergy to contrast media
13. Has any bleeding disorders (tests required if clinical status unknown) or is resistant to aspirin and/or clopidogrel or has any contraindication that precludes antithrombotic treatment
14. Has an allergy to any materials included in the implanted device
15. Has a history of Deep Vein Thrombosis (DVT) or on hormone therapy (eg: HRT)
16. Any serious disease or disorder that in the opinion of the Investigator, could seriously affect ability to participate in the study
17. Does not have a family member/caregiver (or equivalent) who can be present during the consent process and support all study visits
18. Has had any of the following neuropathologies;

    1. Sinus Thrombosis
    2. Venous Hypertension
    3. Hydrocephalus
    4. Bleeding Disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-01-09 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events | 12 month post implant
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
High fidelity and stable signals over 12 months | 36 months
  1. The mean and standard deviation (SD) of first three measurements of impedance values across all 16 channels, excluding flag values, to a maximum of 10 measurements
  2. The mean and SD of noise floor calculated from 2 mins of baseline recording
  3. The mean and SD of signal-to-noise ratio across 3 mins recording of photic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Oxley, Study Director — University of Melbourne and Synchron
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Mitchell P, Lee SCM, Yoo PE, Morokoff A, Sharma RP, Williams DL, MacIsaac C, Howard ME, Irving L, Vrljic I, Williams C, Bush S, Balabanski AH, Drummond KJ, Desmond P, Weber D, Denison T, Mathers S, O'Brien TJ, Mocco J, Grayden DB, Liebeskind DS, Opie NL, Oxley TJ, Campbell BCV. Assessment of Safety of a Fully Implanted Endovascular Brain-Computer Interface for Severe Paralysis in 4 Patients: The Stentrode With Thought-Controlled Digital Switch (SWITCH) Study. JAMA Neurol. 2023 Mar 1;80(3):270-278. doi: 10.1001/jamaneurol.2022.4847. PMID 36622685